CLINICAL TRIAL: NCT02841319
Title: The Effects of Virtual Reality Therapy Compared With Home Exercise Program on Upper Extremity Functions in Children With Hemiplegic Cerebral Palsy: a Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality on Upper Extremity Function in Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sara Asghari Kaleibar, Sara ASGHARI KALEIBAR, MD Resident in the Department of Physical Medicine and Rehabilitation Istanbul Faculty of Medicine, Istanbul University, Istanbul, Turkey, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKaleibar
Record Dates: First submitted 2016-05-21; First posted 2016-07-22 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Cerebral Palsy
Keywords: Virtual reality; Hemiplegic; Cerebral Palsy; upper extremity; hand function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Virtual reality exercises using Hand Tutor for 8 weeks
  Interventions: Other: Virtual Reality Exercises using Hand Tutor
- Control (No Intervention): Home exercises for 8 weeks

INTERVENTIONS:
Other: Virtual Reality Exercises using Hand Tutor — Virtual reality technology is rapidly becoming a popular application for physical rehabilitation and motor control research. The prototype, which includes a built-in movement sensor, allows the user to do controlled exercises as part of a rehabilitation program. The supervised intervention program consists of a forty-minute exercise session three times a week for 8 weeks. In addition, these patients will receive a home exercise program. The patients in the control group will receive only a home exercise program for 8 weeks. The home exercise program consists of different games and exercises such as range of motion, stretch, and strengthening exercises for hand.
  Arms: Intervention

SUMMARY:
The investigators have planned a research on the effects of virtual reality therapy and home exercise program on hand functions in children with hemiplegic cerebral palsy in Istanbul University Istanbul Faculty of Medicine in the Department of Physical Medicine and Rehabilitation. The eligible patients will be randomized into two groups. The patients in intervention group will participate in a computer based virtual reality exercise program for a period of 8 weeks supervised by the investigators. In addition, these patients will receive a home exercise program. The patients in the control group will receive only a home exercise program for 8 weeks. All patients will be evaluated before treatment, immediately after treatment, and 3 months after the end of the treatment.

DETAILED DESCRIPTION:
The current study is a prospective, randomized controlled interventional trial, which will conduct in the Istanbul University Istanbul Faculty of Medicine in 2016. The study was approved by the Ethics Committee in conformity with the Declaration of Helsinki. Prior to data collection, all participants will provide informed consent. By the order of application to the outpatient clinics, the eligible participants will randomly allocated to two groups using the computer-generated random numbers: intervention group (n=17) and control group (n=17). Information on demographic characteristics (age, gender, body mass index, educational level), pre-natal history, parent educational level and past medical history will obtain at baseline assessment. After baseline assessment, the patients in intervention group will participate in a computer based virtual reality exercise program with HandTutor equipment. The supervised intervention program consists of a forty-minute exercise session three times a week for 8 weeks. In addition, these patients will receive a home exercise program. The patients in the control group will receive only a home exercise program for 8 weeks. The home exercise program consists of different games and exercises such as range of motion, stretch, and strengthening exercises for hand. All patients will be evaluated before treatment, immediately after treatment, and 3 months after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with hemiplegic cerebral palsy diagnosed by the specialist
* Active wrist extension ≥ 20 °
* Gross Motor Function Classification System score: 1-2
* Manual Ability Classification System score: 1-3
* The ability to follow simple commands and participate in the task

Exclusion Criteria:

* Contracture in upper limb
* Absence of vision and hearing problems
* Uncontrolled seizure
* Lack of movement in the hemiplegic upper limb
* History of orthopedic surgery (tendon transfer / tendon lengthening) to the affected upper extremity
* Any treatment for upper limb in the last 6 months including BTX-A or orthopedic interventions

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | Within 7 Days
  AHA measures are valid and reliable for children aged between 18 months and 12 years with the diagnosis of unilateral cerebral palsy. It measures how effectively children with unilateral hand dysfunction use their involved hand in collaboration with their uninvolved hand to perform bimanual tasks.The test is administered in two steps. First, a video-recorded play session lasting 10 to 15 minutes is conducted with specific toys from the AHA test kit.Second, the scoring is performed by a review of the video on 22 items by certificated professional. The AHA version 4.4 includes 22 test items each rated on a 4-point scale, with a total raw score range between 22-88 points. The higher score indicating higher ability.

SECONDARY OUTCOMES:
Hand Grip Measurement | Within 7 Days
  Grip strength will measured with BASELINE Dynamometer. The participants will seat and the shoulder is hold in the adducted and minimally internal rotated, elbow flexed at 90 degrees, forearm in natural position and wrist flexed between 0 and 30 degrees (Kg/f).
ABILHAND | Within 7 Days
  ABILHAND-Kids is a measure of manual ability for children with upper limb impairments. The scale measures a person's ability to manage daily activities that require the use of the upper limbs. 21 manual activities perceived by the children parents. Each item is answered on a 3-level scale (impossible, difficult, easy). The Parent is asked to fill in the questionnaire by estimating their child's performance independent of the limb the child actually. The online analysis converts the raw scores into a linear measure of manual ability. ABILHAND-Kids has been validated in cerebral palsy children (age 6-15).
Range of Motion (ROM) | Within 7 Days
  By using the Universal Goniometer, the active and passive ROM will be assessed based on the 360-degrees system in radioulnar pronation and supination, wrist flexion and extension, 2nd to 5th metacarpophalangeal joints
Modified Ashworth Scale (MAS) | Within 7 Days
  One of the methods for measuring muscle spasticity includes manually moving a limb through its ROM to passively stretch specific muscle groups. Modified Ashworth Scale for Grading Spasticity is six-point scale (0-5).
TARDIEU SCALE | Within 7 Days
  Tardieu Scale (TS):
  It assesses the response of the muscle to passive movement of limb in both slow and fast speeds, on the other word it evaluated velocity dependent muscle tonicity. Intensity of muscle reaction (Y) is included six-point scale (0-5)
Pulp Pinch Strength Measurement | Within 7 Days
  Pulp pinch strength is measured by the "JAMAR Hydraulic Pinch Gauge" which evaluates the pinch strength between first and second digits. The participants will seat and the shoulder is hold in the adducted and minimally internal rotated, elbow flexed at 90 degrees, forearm in natural position and wrist flexed between 0 and 30 degrees (Kg/f).

CONTACTS AND LOCATIONS:
Overall Officials: Resa Aydin, MD, Prof, Study Director — Istanbul University Istanbul Faculty of Medicine Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We have no permission to share individual participant data.

REFERENCES:
- [Background] Gabis LV, Tsubary NM, Leon O, Ashkenasi A, Shefer S. Assessment of Abilities and Comorbidities in Children With Cerebral Palsy. J Child Neurol. 2015 Oct;30(12):1640-5. doi: 10.1177/0883073815576792. Epub 2015 Apr 8. PMID 25855688
- [Background] Surveillance of Cerebral Palsy in Europe. Surveillance of cerebral palsy in Europe: a collaboration of cerebral palsy surveys and registers. Surveillance of Cerebral Palsy in Europe (SCPE). Dev Med Child Neurol. 2000 Dec;42(12):816-24. doi: 10.1017/s0012162200001511. PMID 11132255
- [Background] Green D, Schertz M, Gordon AM, Moore A, Schejter Margalit T, Farquharson Y, Ben Bashat D, Weinstein M, Lin JP, Fattal-Valevski A. A multi-site study of functional outcomes following a themed approach to hand-arm bimanual intensive therapy for children with hemiplegia. Dev Med Child Neurol. 2013 Jun;55(6):527-33. doi: 10.1111/dmcn.12113. Epub 2013 Mar 5. PMID 23458353
- [Background] Basu AP, Pearse J, Kelly S, Wisher V, Kisler J. Early intervention to improve hand function in hemiplegic cerebral palsy. Front Neurol. 2015 Jan 6;5:281. doi: 10.3389/fneur.2014.00281. eCollection 2014. PMID 25610423
- [Background] Morris C. Definition and classification of cerebral palsy: a historical perspective. Dev Med Child Neurol Suppl. 2007 Feb;109:3-7. doi: 10.1111/j.1469-8749.2007.tb12609.x. PMID 17370476
- [Background] Meyer-Heim A, van Hedel HJ. Robot-assisted and computer-enhanced therapies for children with cerebral palsy: current state and clinical implementation. Semin Pediatr Neurol. 2013 Jun;20(2):139-45. doi: 10.1016/j.spen.2013.06.006. PMID 23948688
- [Background] Gilliaux M, Renders A, Dispa D, Holvoet D, Sapin J, Dehez B, Detrembleur C, Lejeune TM, Stoquart G. Upper limb robot-assisted therapy in cerebral palsy: a single-blind randomized controlled trial. Neurorehabil Neural Repair. 2015 Feb;29(2):183-92. doi: 10.1177/1545968314541172. Epub 2014 Jul 11. PMID 25015650
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Schiariti V, Klassen AF, Cieza A, Sauve K, O'Donnell M, Armstrong R, Masse LC. Comparing contents of outcome measures in cerebral palsy using the International Classification of Functioning (ICF-CY): a systematic review. Eur J Paediatr Neurol. 2014 Jan;18(1):1-12. doi: 10.1016/j.ejpn.2013.08.001. Epub 2013 Sep 17. PMID 24051208